CLINICAL TRIAL: NCT02038023
Title: Intravaneous Iron(1000 mg Low Molecular Weight Iron Dextran Over 60 Minutes) for Moderate to Severe Iron Deficient Anemia of Pregnancy in Women Intolerant of or Responsive to Oral Iron.
Brief Title: Intravaneous Iron(1000 mg Low Molecular Weight Iron Dextran Over 60 Minutes) for Pregnant Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Auerbach Hematology Oncology Associates P C (Other)
Collaborators: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Intravaneous Iron in Pregnancy; Infed (Other Grant/Funding Number: pharmacosmos)
Record Dates: First submitted 2014-01-09; First posted 2014-01-16 (Estimated); Results first posted 2018-06-28 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-01

CONDITIONS: Pregnancy
Keywords: Iv iron in pregnant women; second and third trimester
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IV iron (Other): Intravaneous iron(1000 mg low molecular weight iron dextran over 60 minutes) for moderate to severe iron deficient anemia of pregnancy in women intolerant of or unresponsive to oral iron.
  Interventions: Drug: Intravaneous iron(low molecular weight iron dextran)

INTERVENTIONS:
Drug: Intravaneous iron(low molecular weight iron dextran) — 1000 mg of Iron dextran administered over one hour
  Other Names: Iron Dextran(InFed)

SUMMARY:
To determine the percentage of women who achieve anemia correction after a single dose of 1000mg of low molecular weight iron dextran(infed).

DETAILED DESCRIPTION:
To determine the percentage of women who achieve anemia correction after a single dose of 1000mg of low molecular weight iron dextran(infed).

To determine whether IV iron supplementation has a higher satisfaction with treatment as compared to oral supplementation in a population previously intolerant of or unresponsive to oral iron.

To evaluate the safety of IV low molecular weight iron dextran in pregnant women.

To assess maternal and fetal outcomes-preterm delivery, low birth weight deliveries, ER visits and hospitalizations related to preterm labor, preterm contractions, ante-partum and post-partum transfusions, maternal hemoglobin at post-partum visit after IV iron supplementation groups.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women intolerable to oral iron. hbg <10.9 g/dl during second or third trimester.

Exclusion Criteria:

* known sensitivity to IV iron. hemoglobinopathies. hemolytic anemia. women who have received or will receive blood transfusions. women with significant vaginal bleeding(>200 cc blood loss)prior to delivery. women with documented history of allergy to more than one class of drug clinically significant anemia requiring therapy in the opinion of the obstetrician, in the first trimester.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Auerbach, MD, Principal Investigator — Auerbach Hematology Oncology
Locations (1):
- Auerbach Hematology Oncology Assoc, Baltimore, Maryland, United States

REFERENCES:
- [Result] Auerbach M, James SE, Nicoletti M, Lenowitz S, London N, Bahrain HF, Derman R, Smith S. Results of the First American Prospective Study of Intravenous Iron in Oral Iron-Intolerant Iron-Deficient Gravidas. Am J Med. 2017 Dec;130(12):1402-1407. doi: 10.1016/j.amjmed.2017.06.025. Epub 2017 Jul 21. PMID 28739199

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Standard referrals from obstetricians and gynecologists
Pre-assignment Details: Oral iron intolerance plus iron deficiency anemia as defined by a serum ferritin of <20 ng/mL or transferrin saturation of <19% in the 2nd or 3rd trimester plus the ACOG guidelines of <10/.5 g/dL and 11.0 g/dl respectively. 73/74 enrolled received the planned dose.
Period: Overall Study
Arm/Group | IV Iron
Started | 74
Completed | 73
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Iron deficient gravidas in 2nd and 3rd trimesters
Groups:
- Intravenous Iron: As oral iron intolerant iron deficient 2nd and 3rd trimester gravidas defined by a ferritin of <20 ng/mL and TSAT ,19%. All were anemic by ACOG criteria of Hb <10.5 g/dL in 2nd trimester or, 11g/dL in 3rd, who received 1000 mg IV low molecular weight iron dextran in one hour
Arm/Group | Intravenous Iron
Number analyzed (Participants) | 74
Age, Continuous [Mean (Full Range); unit: years] | 24 [18 to 42]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  All female | 74
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 74
Pretreatment Hb [Mean (Standard Deviation); unit: g/dL] | 9.65 (0.70)
Iron Deficient Pregnant Gravidas [Count of Participants; unit: Participants] | 74
Serum ferritin [Mean (Standard Deviation); unit: ng/mL] | 14.53 (24.61)
Percent Transferrin Saturation [Mean (Standard Deviation); unit: percent saturation (Fe/TIBC)] | 11.72 (9.14)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Women Who Achieve Anemia Correction After a Single Dose of 1000mg of Low Molecular Weight Iron Dextran(INfeD).
Time Frame: 4 weeks after infusion or post-partum
Population: Of the 73 who received the infusion, 5 were lost to followup and 8 did not return for 4-week posttreatment bloodwork. Pretreatment (initial) and 4-week posttreatment laboratory studies are available for 60
Measure: Count of Participants; unit: Participants
Groups:
- Iron Deficient Gravidas: This has been described twice before. Iron deficient pregnant women in the 2nd and 3rd trimester
Arm/Group | Iron Deficient Gravidas
Number analyzed (Participants) | 60
Participants
  Improvement of > or equal to 1 g/dL | 35
  Improvement of > or equal to 2 g/dL | 11

2. Secondary Outcome: Serum Ferritin
Time Frame: 4 weeks post infusion or post-partum
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Intravenous Iron: As oral iron intolerant iron deficient 2nd and 3rd trimester gravidas defined by a ferritin of <20 ng/mL and TSAT, 19%. All were anemic by ACOG criteria of Hb <10.5 g/dL in 2nd trimester or, 11g/dL in 3rd, who received 1000 mg IV low molecular weight iron dextran in one hour
Arm/Group | Intravenous Iron
Number analyzed (Participants) | 60
ng/mL | 126.29 (88.48)

3. Secondary Outcome: Percent Transferrin Saturation
Time Frame: 4 weeks post infusion or post-partum
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent saturation (Fe/TIBC)
Arm/Group | Iron Deficient Gravidas
Number analyzed (Participants) | 60
percent saturation (Fe/TIBC) | 22.64 (12.14)

4. Secondary Outcome: Safety as Measured by Number of Adverse Events
Description: To evaluate the safety of IV low molecular weight iron dextran in pregnant women. Also to asses maternal and fetal outcomes-preterm delivery, low-birth weight deliveries, ER visits and hospitalizations related to preterm labor, preterm contractions, ante-partum and post partum transfusions, maternal hemoglobin at post-partum visit after IV iron supplementation groups. A questionaire with a list of symptoms to include nausea, dizziness, hypotension, edema, headache, abdominal pain, chest pain, cough, itching, fever, back pain, muscle cramps and rash are asked immediately after administration and phone calls at 24, 48 hours and 7 days.
Time Frame: 4 weeks after infusion and 4 weeks post-partum
Measure: Number; unit: minor adverse events
Groups:
- Only One Group[: Post treatment hemoglobin in 73/74 gravidas
Arm/Group | Only One Group[
Number analyzed (Participants) | 74
minor adverse events | 6

ADVERSE EVENTS:
Arm/Group | IV Iron
Serious Adverse Events (participants affected / at risk) | 0/74
Other Adverse Events (participants affected / at risk) | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes